CLINICAL TRIAL: NCT03858491
Title: Pharmacokinetic Boosting of Osimertinib in Patients With Non-small Cell Lung Cancer.
Brief Title: Pharmacokinetic Boosting of Osimertinib
Acronym: OSIBOOST
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Academisch Ziekenhuis Maastricht (Other)
Collaborators: The Netherlands Cancer Institute (Other); ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Principal Investigator, Ard van Veelen, Researcher, Academisch Ziekenhuis Maastricht
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-004290-28
Record Dates: First submitted 2019-02-26; First posted 2019-02-28 (Actual); Last update posted 2022-09-26 (Actual); Status verified 2022-09

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Osimertinib; Cobicistat; Pharmacokinetic boosting
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Cobicistat

STUDY DESIGN:
Intervention Model Description: In this study a group of patients will receive cobicistat as add-on on their regular treatment with osimertinib. All patients experience low osimertinib trough concentration levels when treated with the regular osimertinib dose (80 mg per day).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cobicistat (Experimental): Cobicistat will serve as experimental drugs, and will be added to the regular treatment with osimertinib. Combination-treatment will be started at 150 milligram cobicistat, and can be increased to a maximum daily dose of 600 milligram cobicistat (four times 150 milligram).
  Interventions: Drug: Cobicistat

INTERVENTIONS:
Drug: Cobicistat — Cobicistat will be added to the treatment with osimertinib. The initial dose will be 150 mg cobicistat, which equals the dose used in the treatment of HIV-infected patients. If this dose is well tolerated and the increase in exposure of osimertinib is not sufficient, the dose of cobicistat will gradually be escalated to 600 mg per day (150 mg cobicistat, four times per day).
  Other Names: Tybost

SUMMARY:
The main objective of this study is to evaluate if systemic exposure of osimertinib (i.e. AUC) is increased when osimertinib is co-administered with cobicistat in patients with relatively low plasma trough concentration while receiving the standard osimertinib dose.

DETAILED DESCRIPTION:
Osimertinib is a new targeted agent registered for the treatment of patients with EGFR-mutated NSCLC. However, the costs of those new treatments are extremely high. Osimertinib is mainly metabolized by CYP3A4, and partially by CYP3A5. Combination of osimertinib with a strong CYP3A4-inhibitor may result in a smaller first-pass effect and a decreased clearance of osimertinib, thereby increasing the exposure to osimertinib.

Cobicistat is a strong CYP3A4-inhibitor, this mechanism may be used to boost osimertinib, as is done for other drugs, mainly drugs used to treat HIV-infected patients.

Using this personalized treatment approach and combining the concepts of therapeutic drug monitoring (TDM) and pharmacokinetic boosting, osimertinib therapy could become much more cost-effective. By reducing the necessary dose of osimertinib, this strategy may ultimately result in a significant reduction in drug costs, as the additional expenditure for the CYP3A4 inhibitor and blood sample analysis are negligible compared to the price of osimertinib.

ELIGIBILITY:
Inclusion Criteria:

* Patients with EGFR-mutated NSCLC receiving standard treatment with osimertinib for at least 2 months (steady state), without any signs of disease progression, or during treatment beyond progression, if treatment continuation is expected for multiple months. After anticipated EMA approval of osimertinib adjuvant therapy, patients on adjuvant osimertinib treatment may also participate on the following conditions; If they are receiving standard treatment with osimertinib for at least 2 months (steady state), and if treatment will be continued for a longer period than necessary for participation in the OSIBOOST trial.
* Age ≥ 18 years
* WHO performance status ≤ 2.
* Able and willing to give written informed consent.
* Able and willing to undergo blood sampling for pharmacokinetic analysis.
* Patients with osimertinib plasma trough concentration below 195 ng/mL. Plasma trough concentration of osimertinib will be determined in another study (METC MUMC: 2018-0800).

Exclusion Criteria:

* Any concurrent medication that is known to strongly inhibit or induce CYP3A4.
* Any concurrent medication that is primarily metabolized by CYP3A4 with a narrow therapeutic window.
* Impairment of gastrointestinal function that may alter the absorption of osimertinib or cobicistat (e.g. ulcerative disease, uncontrolled nausea or vomiting, malabsorption syndrome, small bowel resection).
* Refusing to refrain from consuming CYP3A4 influencing products, e.g. grapefruit(juice), St. John's wort.
* Pregnancy or breast feeding
* Child-Pugh score class C, chronic liver disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Osimertinib AUC | Three weeks
  Exposure to osimertinib will be measured at the start of the study and after three weeks of treatment with cobicistat. This will be done by measuring the concentration of osimertinib four times during the day (pre-dose and two, four and eight hour post-dose), which will be used to calculate the AUC of osimertinib.

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0. | Three weeks
  The safety of the combination therapy will be evaluated and scored using NCI CTCAE v4.0. The investigators will evaluate the number of patients that experience treatment-related adverse events. Additionally, the investigators will describe the adverse events which are most common in the lung cancer patients.
  Participants will be asked to keep up a patient diary with problems they have experienced during the study.
Cmax of osimertinib | Three weeks
  The maximum plasma of osimertinib will be determined

CONTACTS AND LOCATIONS:
Overall Officials: Sander Croes, MSc, PhD, Study Director — Maastricht University Medical Centre+ (MUMC+)
Locations (2):
- Netherlands (2):
  - Maastricht University Medical Centre, Maastricht, Limburg
  - Antoni van Leeuwenhoek hospital, Amsterdam, North Holland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Soria JC, Ohe Y, Vansteenkiste J, Reungwetwattana T, Chewaskulyong B, Lee KH, Dechaphunkul A, Imamura F, Nogami N, Kurata T, Okamoto I, Zhou C, Cho BC, Cheng Y, Cho EK, Voon PJ, Planchard D, Su WC, Gray JE, Lee SM, Hodge R, Marotti M, Rukazenkov Y, Ramalingam SS; FLAURA Investigators. Osimertinib in Untreated EGFR-Mutated Advanced Non-Small-Cell Lung Cancer. N Engl J Med. 2018 Jan 11;378(2):113-125. doi: 10.1056/NEJMoa1713137. Epub 2017 Nov 18. PMID 29151359
- [Result] Mok TS, Wu Y-L, Ahn M-J, Garassino MC, Kim HR, Ramalingam SS, Shepherd FA, He Y, Akamatsu H, Theelen WS, Lee CK, Sebastian M, Templeton A, Mann H, Marotti M, Ghiorghiu S, Papadimitrakopoulou VA; AURA3 Investigators. Osimertinib or Platinum-Pemetrexed in EGFR T790M-Positive Lung Cancer. N Engl J Med. 2017 Feb 16;376(7):629-640. doi: 10.1056/NEJMoa1612674. Epub 2016 Dec 6. PMID 27959700
- [Result] Lubberman FJE, van Erp NP, Ter Heine R, van Herpen CML. Boosting axitinib exposure with a CYP3A4 inhibitor, making axitinib treatment personal. Acta Oncol. 2017 Sep;56(9):1238-1240. doi: 10.1080/0284186X.2017.1311024. Epub 2017 Apr 7. No abstract available. PMID 28388255
- [Derived] Westra N, Kruithof PD, Croes S, van Geel RMJM, Hendriks LEL, Touw DJ, Oude Munnink TH, Mian P. Systematic Evaluation of Osimertinib Population Pharmacokinetic Models in a Cohort of Dutch Adults with Non-Small Cell Lung Cancer. Eur J Drug Metab Pharmacokinet. 2024 Jul;49(4):517-526. doi: 10.1007/s13318-024-00904-5. Epub 2024 Jun 15. PMID 38878145
- [Derived] van Veelen A, Gulikers J, Hendriks LEL, Dursun S, Ippel J, Smit EF, Dingemans AC, van Geel R, Croes S. Pharmacokinetic boosting of osimertinib with cobicistat in patients with non-small cell lung cancer: The OSIBOOST trial. Lung Cancer. 2022 Sep;171:97-102. doi: 10.1016/j.lungcan.2022.07.012. Epub 2022 Jul 25. PMID 35933915